CLINICAL TRIAL: NCT01149330
Title: Evaluation of Efficacy and Safety of Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel in the Treatment of Acne Vulgaris
Brief Title: Evaluation of Efficacy and Safety of Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel in the Treatment of Acne Vulgaris
Acronym: Estudo Epiduo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma Brasil Ltda. (Industry)
Responsible Party: Alessandra Nogueira, MD, Galderma Brasil Ltda.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR.10.001
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Acne Vulgaris
Keywords: Adapalene; Benzoyl Peroxide; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adapalene-BPO Gel (Experimental)
  Interventions: Drug: Adapalene-BPO Gel

INTERVENTIONS:
Drug: Adapalene-BPO Gel — Apply 1 gram of the investigational drug every night on whole face.

SUMMARY:
The purpose of this study is to demonstrate the efficacy of Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel in the treatment of acne vulgaris. The safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Subjects, aged 12 to 35 years inclusive, with moderate to severe facial acne vulgaris (described scale score of 3 or 4),
* Subjects with a minimum of 20 and a maximum of 50 Inflammatory Lesions (papules and pustules) on the face, excluding the nose,
* Subjects with a minimum of 30 and a maximum of 100 Non-Inflammatory Lesions (open comedones and closed comedones) on the face, excluding the nose,
* Female Subjects of childbearing potential with a negative urine pregnancy test at the Baseline visit and must practice a highly effective method of contraception during the study: oral/systemic [injectable, patch…] contraception (must have been on a stable dose for 3 months prior to study entry), Intrauterine Device, strict abstinence, condoms, diaphragms, sponge, spermicides or partner had a vasectomy,
* Females of non-childbearing potential, i.e., premenses, post-menopausal (absence of menstrual bleeding for 2 years), hysterectomy, bilateral tubal ligation, or bilateral ovariectomy, secondary infertility and sterility are not required to have a UPT at the beginning of the study,
* Subjects have to read and sign the approved the Informed Consent form prior to any participation in the study. Subjects under the majority must sign an assent-to-participate form to participate in the study and they must have one parent or guardian read and sign the Informed Consent form prior to any study related procedure,
* Subjects willing and capable of cooperating to the extend and degree required by the protocol.

Exclusion Criteria:

* Subjects who have participated in another investigational drug or device research study within 30 days of enrollment,
* Female Subjects who are pregnant, nursing or planning a pregnancy during the study,
* Subjects with more than 1 nodule or cyst on the face
* Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.),
* Subjects with known or suspected allergy to one of the investigational products (see package insert and/or investigator brochure),
* Subjects who have pathological conditions photosensitive porphyria, SLE, LED, solar polymorphous eruption, actinic prurigo, solar urticaria, etc.
* Subjects with a beard or other facial hair that might interfere with study assessments,
* Subjects who foresee intensive UV exposure during the study (mountain sports, UV radiation, sunbathing, etc...)
* Female subjects with a history of hormonal changes.
* Subjects with skin condition or disease requiring topical or systemic therapy, which interferes with the investigational product or that may directly affect the evaluation criteria:

  * Topical treatment for acne in the past two weeks.
  * Anti-inflammatory topic in the last two weeks.
  * Use of topical corticosteroids on the face in the last four weeks.
  * Anti-inflammatory systemic (hormonal or not) in the last four weeks.
  * Use of systemic corticosteroids in the last four weeks.
  * Systemic antibiotics in the last four weeks (excluding penicillins).
  * Systemic retinoids in the last six months.
  * Other systemic anti-acne the last four weeks.
  * Anticonceptional oral used exclusively for the control of acne in the past six months.
  * Cosmetic procedures such as facials, peels, exfoliation, extraction of comedones, application of LED, laser or pulsed light in the last two weeks.
  * Cosmetic procedures such as PDT in the last four weeks.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation | Week 12
  Changing from Baseline in Total Lesion count (Non-Inflammatory and Inflammatory lesions) in Week 12.

SECONDARY OUTCOMES:
Secondary efficacy evaluation | Week 1
  Changing from Baseline in Total Lesion count (Non-Inflammatory and Inflammatory lesions) in Week 1.
Secondary efficacy evaluation | Week 2
  Changing from Baseline in Total Lesion count (Non-Inflammatory and Inflammatory lesions) in Week 2.
Changing from Baseline in Total Lesion count (Non-Inflammatory and Inflammatory lesions) in Week 2. Secondary efficacy evaluation | Week 4
  Changing from Baseline in Total Lesion count (Non-Inflammatory and Inflammatory lesions) in Week 4.
Secondary efficacy evaluation | Week 8
  Changing from Baseline in Total Lesion count (Non-Inflammatory and Inflammatory lesions) in Week 8.
Secondary efficacy evaluation | Week 12
  Changing from Baseline in Total Lesion count (Non-Inflammatory and Inflammatory lesions) in Week 12.
  Assessment of the severity of facial acne. Evaluation of global improvement at study completion. Assessment of improvement and patient satisfaction.
Safety evaluation | Week 1
  Local tolerability scores - Erythema, Scaling, Dryness, Stinging/Burning at each study visit.
Safety evaluation | Week 2
  Local tolerability scores - Erythema, Scaling, Dryness, Stinging/Burning at each study visit.
Safety evaluation | Week 4
  Local tolerability scores - Erythema, Scaling, Dryness, Stinging/Burning at each study visit.
Safety evaluation | week 8
  Local tolerability scores - Erythema, Scaling, Dryness, Stinging/Burning at each study visit.
Safety evaluation | Week 12
  Local tolerability scores - Erythema, Scaling, Dryness, Stinging/Burning at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra T Nogueira, MD, Study Director — Galderma Brasil Ltda.
Locations (6):
- Brazil (6):
  - Serviço de Dermatologia do Ambulatório Magalhães Neto do Complexo HUPES - Universidade Federal da Bahia, Salvador, Estado de Bahia
  - Instituo da Pele, Goiânia, Goiás
  - Hospital De Clínicas - Universidade Federal do Paraná, Curitiba, Paraná
  - Instituto de Dermatologia e Estética do Brasil Ltda., Rio de Janeiro, Rio de Janeiro
  - KOLderma Instituto de Pesquisa Clínica Ltda, Campinas, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual, São Paulo, São Paulo